CLINICAL TRIAL: NCT04725097
Title: Rapid Throughput Screening for Human COVID-19 Infection: A ECG Study
Brief Title: A Study to Evaluate Rapid Throughput Screening for Human COVID-19 Infection
Status: Terminated | Type: Observational
Why Stopped: Interim analysis indicated adaptions may be required.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elie F. Berbari, Principal Investigator, Mayo Clinic
Other Study IDs: 20-011415
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the ability of an artificial intelligence smartphone-enabled point of care ECG to detect COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females age 18 or greater.
* Undergoing COVID-19 testing by PCR.
* Willing and able to provide informed consent.
* Pregnant females (minimal risk study, no risk from ECG).

Exclusion Criteria:

- Unwilling or unable to provide informed consent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Detection of COVID-19 when compared to a PCR test in asymptomatic patients.
Sampling Method: Probability Sample
Enrollment: 2821 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
COVID 19 Detection | One time screening within 4 hours of PCR test
  Determine the safety and feasibility of the POC AI-ECG's ability to detect active SARS-Cov-2 infection in humans.

CONTACTS AND LOCATIONS:
Overall Officials: Elie F Berbari, MD, Principal Investigator — Mayo Clinic
Locations (10):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - LSUHSC Shreveport, Shreveport, Louisiana
  - Henry Ford Health System, West Bloomfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack Meridian Health, Hackensack, New Jersey
- India (2):
  - Sri Jayadeva, Bengaluru, Karnataka
  - King Edward Memorial Hospital, Mumbai, Maharashtra
- Gregorio Marañon Hospital, Madrid, Spain
- Imperial College, London, England, United Kingdom

REFERENCES:
- [Derived] Adedinsewo D, Dugan J, Johnson PW, Douglass EJ, Morales-Lara AC, Parkulo MA, Ting HH, Cooper LT, Scott LR, Valverde AM, Padmanabhan D, Peters NS, Bachtiger P, Kelshiker M, Fernandez-Aviles F, Atienza F, Glotzer TV, Lahiri MK, Dominic P, Attia ZI, Kapa S, Noseworthy PA, Pereira NL, Cruz J, Berbari EF, Carter RE, Friedman PA. RApid Throughput Screening for Asymptomatic COVID-19 Infection With an Electrocardiogram: A Prospective Observational Study. Mayo Clin Proc Digit Health. 2023 Sep 16;1(4):455-466. doi: 10.1016/j.mcpdig.2023.07.007. eCollection 2023 Dec. PMID 40206301
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials